CLINICAL TRIAL: NCT07135934
Title: Evaluation of the Effects of Single Sodium Bicarbonate Supplementation on Finswimming Performance of National Level Finswimmers: A Randomized, Double-Blind, Placebo-Controlled Crossover Study
Brief Title: Effects of Single Sodium Bicarbonate Supplementation on National-Level Finswimming Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Palacky University (Other)
Responsible Party: Principal Investigator, Tomáš Michalica, Principal Investigator, Doctoral Researcher and Assistant Lecturer, Faculty of Physical Culture, Palacký University Olomouc, Palacky University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: FTK_2024_002
Record Dates: First submitted 2025-08-01; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Sport Performance; Acid Base Imbalance; Ergogenic Support; Sodium Bicarbonate; Water Sports; Biomechanics
Keywords: Sodium Bicarbonate; Stroke Rate; Finswimming; Stroke Length; Athletes; Biomechanics; Gastrointestinal Discomfort; Rate of Perceived Exertion
MeSH Terms: conditions — Acid-Base Imbalance | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator (Placebo Comparator): Placebo: Food-grade starch Participants will ingest 300 mg·kg-¹ body mass of food-grade starch encapsulated in gelatin capsules 60-90 minutes prior to the simulated 200 m Bi-Fins race.
  Dietary Supplement: Placebo Gelatin capsules filled with food-grade starch, indistinguishable in appearance from sodium bicarbonate capsules. Water is consumed ad libitum during ingestion.
  Other Names: Placebo Capsules
  Interventions: Dietary Supplement: Placebo
- Sodium Bicarbonate (NaHCO₃) (Experimental): Sodium Bicarbonate: NaHCO₃ Participants will ingest 300 mg·kg-¹ body mass of sodium bicarbonate encapsulated in gelatin capsules 60-90 minutes prior to the simulated 200 m Bi-Fins race.
  Dietary Supplement: Sodium Bicarbonate Gelatin capsules containing sodium bicarbonate (NaHCO₃), matched in appearance, weight, and texture to placebo. Water is consumed ad libitum during ingestion.
  Other Names: NaHCO₃ Capsules
  Interventions: Dietary Supplement: Sodium Bicarbonate (NaHCO3)

INTERVENTIONS:
Dietary Supplement: Sodium Bicarbonate (NaHCO3) — Gelatin capsules each containing 1g sodium bicarbonate (NaHCO₃)
  Arms: Sodium Bicarbonate (NaHCO₃)
Dietary Supplement: Placebo — Gelatin capsules each containing 1g food-grade starch
  Arms: Placebo Comparator

SUMMARY:
This randomized, double-blind, placebo-controlled crossover trial will investigate the acute effects of sodium bicarbonate supplementation on performance, stroke biomechanics, and selected physiological and perceptual responses during a simulated 200-meter Bi-Fins race in elite finswimmers.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, crossover study will examine the effects of sodium bicarbonate (NaHCO₃) supplementation on simulated finswimming performance and associated biomechanical, physiological, and perceptual responses in national-level finswimmers. Twenty participants, all active members of the Czech junior or senior national team, will complete three test sessions separated by a 48-hour recovery period without training sessions.

The first session will serve as a control with no intervention, while the second and third will involve ingestion of either sodium bicarbonate (NaHCO₃; 300 mg·kg-¹) or placebo (food-grade starch), administered in a randomized, counterbalanced order. The capsules will be indistinguishable in appearance, weight, and texture. Allocation concealment will be ensured: only a designated medical professional overseeing the health and safety of the participants will have access to the randomization codes. Neither the participants nor the investigators will be aware of the supplement condition during testing.

All sessions will be conducted under standardized conditions in a 25-meter indoor swimming pool (Aplikační centrum BALUO, Palacký University Olomouc) and will include a standardized warm-up followed by a 200-meter Bi-Fins time trial.

Blood samples for acid-base balance assessment will be collected at four time points: baseline (10 minutes before warm-up), 10 minutes after warm-up, 5 minutes before race start, and 3 minutes post-exercise. From these samples, variability in acid-base balance will be assessed, specifically using actual base excess (ABE; mmol/L), blood hydrogen ion concentration (pH; unitless), and bicarbonate concentration (HCO₃-; mmol/L). Blood lactate concentration (mmol/L) will be measured at two time points only: baseline (10 minutes before warm-up) and 3 minutes post-exercise.

Subjective perceptual responses will include:

1. rate of perceived exertion (RPE) using the Borg Category Ratio 1-10 scale, assessed immediately after the race, where higher scores indicate greater exertion;
2. gastrointestinal discomfort using the Borg Category Ratio 1-10 scale, assessed approximately 5 minutes before the race to avoid performance bias, where higher scores indicate worse discomfort; and
3. delayed-onset muscle soreness (DOMS) using a 10-centimeter visual analog scale (VAS; 0 cm = no soreness, 10 cm = extreme soreness) for both upper and lower limbs, where higher scores indicate greater soreness.

Stroke mechanics - stroke rate (SR; cycles/min) and stroke length (SL; meters/cycle) - will be analyzed from video recordings of the 200-meter trials.

The study will follow the Consolidated Standards of Reporting Trials (CONSORT) guidelines for crossover trials and has been approved by the Ethics Committee of the Faculty of Physical Culture, Palacký University Olomouc (Ref. No. 2/2024).

Statistical analysis will include repeated-measures analysis of variance (ANOVA) to compare conditions and time points. In case of violation of assumptions, appropriate corrections or non-parametric alternatives will be applied. Descriptive statistics, effect sizes (partial eta-squared, Cohen's d), and correlation coefficients (Pearson's r) will be used to support the interpretation of results. Data will be processed using International Business Machines Statistical Package for the Social Sciences (IBM SPSS) software and Microsoft Excel.

ELIGIBILITY:
Inclusion Criteria:

1. Member of a wider national selection in finswimming (junior or senior level)
2. Regular participation in competitive finswimming training (≥4 sessions per week)
3. Age between 15 and 30 years
4. Absence of chronic illness or injury
5. No use of medications or dietary supplements during the study period
6. Signed informed consent (for minors, also signed by a legal guardian)

Exclusion Criteria:

1. History of gastrointestinal disorders affecting supplement tolerance
2. Presence of cardiovascular, metabolic, or musculoskeletal disorders
3. Current illness or acute infection
4. Regular use of substances that may interfere with acid-base balance
5. Refusal to comply with pre-test restrictions (e.g., 48 hours without training)

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-08-17 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Stroke rate (SR; cycles/min) | Measured from video analysis of the 200-m Bi-Fins trial; final values reported at race completion on Day 1, Day 3, and Day 5.
  Calculated from video analysis to determine the number of stroke cycles per minute.
Total race time (seconds) | Measured from video analysis of the 200-m Bi-Fins trial; final values reported at race completion on Day 1, Day 3, and Day 5.
  Total time to complete the 200-meter Bi-Fins time trial, measured using an electronic timing system. Lower values indicate better performance.
Stroke length (SL; meters/cycle) | Measured from video analysis of the 200-m Bi-Fins trial; final values reported at race completion on Day 1, Day 3, and Day 5.
  Calculated from video analysis to determine the average distance traveled per stroke cycle.

SECONDARY OUTCOMES:
Underwater distance (meters) | Measured from video analysis of the 200-m Bi-Fins trial; final values reported at race completion on Day 1, Day 3, and Day 5.
  Distance traveled underwater after the start and turns, measured from video footage of the 200-meter Bi-Fins time trial. Greater values indicate a longer underwater phase.
Blood lactate concentration (mmol/L) | Baseline (10 minutes before warm-up) and 3 minutes post-exercise on each testing day
  Measured from capillary blood samples to assess anaerobic metabolism. Higher values indicate greater lactate accumulation.
Actual base excess (ABE; mmol/L) | Baseline (10 minutes before warm-up), 10 minutes after warm-up, 5 minutes before race start, and 3 minutes post-exercise on each testing day
  Measured from capillary blood samples to assess buffering capacity. More negative values indicate greater metabolic acidosis.
Blood bicarbonate concentration (HCO₃-; mmol/L) | Baseline (10 minutes before warm-up), 10 minutes after warm-up, 5 minutes before race start, and 3 minutes post-exercise on each testing day
  Measured from capillary blood samples to assess bicarbonate availability for acid buffering. Lower values indicate reduced buffering capacity.
Rate of Perceived Exertion (RPE; score on Borg Category Ratio 1-10 scale) | Immediately post-exercise on each testing day
  The Borg Category Ratio 1-10 scale ranges from 1 (no exertion at all) to 10 (maximal exertion). Higher scores indicate greater exertion.
Gastrointestinal discomfort (score on Borg Category Ratio 1-10 scale) | Approximately 5 minutes before race start on each testing day
  The Borg Category Ratio 1-10 scale ranges from 1 (no discomfort) to 10 (severe discomfort). Higher scores indicate worse discomfort.
Delayed-onset muscle soreness (DOMS; score on 10-centimeter visual analog scale) | Immediately post-exercise on each testing day
  The visual analog scale (VAS) ranges from 0 cm (no soreness) to 10 cm (extreme soreness). Higher scores indicate greater soreness.
Underwater time (seconds) | Measured from video analysis of the 200-m Bi-Fins trial; final values reported at race completion on Day 1, Day 3, and Day 5.
  Time spent underwater after the start and turns, measured from video footage of the 200-meter Bi-Fins time trial. Greater values indicate a longer underwater phase.
Underwater velocity (meters/second) | Measured from video analysis of the 200-m Bi-Fins trial; final values reported at race completion on Day 1, Day 3, and Day 5.
  Average velocity during the underwater phase after the start and turns, measured from video footage of the 200-meter Bi-Fins time trial. Higher values indicate faster underwater performance.
Blood hydrogen ion concentration (pH; unitless) | Baseline (10 minutes before warm-up), 10 minutes after warm-up, 5 minutes before race start, and 3 minutes post-exercise on each testing day
  Measured from capillary blood samples to assess acid-base balance. Higher or lower values indicate changes in blood acidity.

CONTACTS AND LOCATIONS:
Overall Officials: Tomáš Michalica, Mgr., Principal Investigator — Palacký University, Faculty of Physical Culture
Locations (1):
- Palacký University, Faculty of Physical Culture, Olomouc, Olomoucký kraj, Czechia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Time Frame: Beginning 1 year after the publication of results with no end date.